CLINICAL TRIAL: NCT02313298
Title: A Phase II Trial of Prostate Stereotactic Radiotherapy
Brief Title: Stereotactic Body Radiotherapy for Organ Confined Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCS DRO SBRT
Record Dates: First submitted 2014-12-07; First posted 2014-12-10 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic Body Radiotherapy (Experimental): An extreme hypofractionated regimen of 36.25Gy in 5 fractions over 10-11 days
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — IMRT or similar techniques that use inverse treatment planning

SUMMARY:
A single arm phase II study of SBRT for prostate cancer to primarily assess acute and late toxicity and secondarily PSA outcomes and quality of life measurements of an extreme hypofractionated regimen of 36.25Gy in 5 fractions over 10-11 days.

DETAILED DESCRIPTION:
This is a single arm phase II study of SBRT for prostate cancer to primarily assess acute and late toxicity and secondarily PSA outcomes and quality of life measurements of an extreme hypofractionated regimen of 36.25Gy in 5 fractions over 10-11 days. The radiation therapy is to be delivered using intensity modulated radiotherapy (IMRT) with the aid of volumetric image guidance to ensure accuracy. Toxicity will be measured at preset intervals, as will HRQOL parameters using the Expanded Prostate Index Composite (EPIC) questionaire which focuses on bowel, urinary, sexual and hormonal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate
* History/physical examination with digital rectal examination of the prostate within 60 days prior to registration
* Histological evaluation of prostate biopsy with assignment of a Gleason score to the biopsy material; Gleason scores 2-7
* Clinical stage T1-2b (DRE) (AJCC 7th edition) within 90 days of registration
* PSA < 20 ng/mL within 60 days prior to registration. PSA should not be obtained within 10 days after prostate biopsy. (Every effort should be made to obtain all serum PSA values obtained in the 1 year prior to treatment to allow for calculation of PSA kinetics.)
* Not more than one intermediate risk factor (T2b/GS7/PSA 10-20)
* Zubrod Performance Status 0-1 within 60 days prior to registration
* Age ≥ 21
* Patient must be able to provide study-specific informed consent prior to study entry.
* Willingness and ability to complete the Expanded Prostate Cancer Index Composite (EPIC) questionnaire

Exclusion Criteria:

* Prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease free for a minimum of 5 years. (For example, carcinoma of the oral cavity is permissible; however, patients with prior history of bladder cancer are not allowed)
* T-stage ≥ T2c on staging MRI
* Evidence of distant metastases
* Regional lymph node involvement
* Previous radical surgery (prostatectomy), cryosurgery, or HIFU for prostate cancer
* Previous pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy
* Previous hormonal therapy, such as LHRH agonists (e.g., goserelin, leuprolide) or LHRH antagonists (e.g., degarelix), anti-androgens (e.g., flutamide, bicalutamide), estrogens (e.g., DES), or surgical castration (orchiectomy)
* Use of finasteride within 30 days prior to registration. PSA should not be obtained prior to 30 days after stopping finasteride.
* Use of dutasteride within 90 days prior to registration. PSA should not be obtained prior to 90 days after stopping dutasteride.
* Previous or concurrent cytotoxic chemotherapy for prostate cancer
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol. (Patients on Coumadin or other blood thinning agents are eligible for this study.)
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2018-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The rate of late severe GI and GU toxicities | 2 years

SECONDARY OUTCOMES:
The rate of late severe GI and GU toxicities | 1 and 5 years
The rate of acute severe GI and GU toxicities | 1, 2 and 5 years
PSA failure-free survival | 1, 2 and 5 years
Disease-free survival (DFS) | 1, 2 and 5 years
Time to local progression | 1, 2 and 5 years
Time to distant and/or regional failure | 1, 2 and 5 years
Disease-specific survival | 1, 2 and 5 years
Freedom from biochemical recurrence (FFBR) | 1, 2 and 5 years
Overall survival (OS) | 1, 2 and 5 years
The change in quality of life outcomes from baseline | 1, 2 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Melvin LK Chua, Study Director — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore